CLINICAL TRIAL: NCT05828797
Title: Evaluation of Shoulder Region With Share-Wave Ultrasound Elastography in Patients With Hemiplegia
Brief Title: Elastography in Patients With Hemiplegia
Status: Recruiting | Type: Observational
Sponsor: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Veysel Delen, MD, MD, Harran University
Other Study IDs: HRU
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Hemiplegia; Elastography; Shoulder; Muscles
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Shoulder elastography on the hemiplegic side of patients: Patients over the age of 18 who apply to our clinic and have hemiplegia complaints will be evaluated. Patients' age, gender, occupation, habits, disease duration, upper extremity with complaints, dominant upper extremity, additional disease, weight and height values will be recorded. In the physical medicine and rehabilitation department examination of the patients, the patients will be evaluated with the brunnstrom staging used in hemiplegic patients. The elastography of the shoulder on the side with hemiplegia and the elastography of the shoulder on the side without complaints will be examined. Thus, the patient's side with the complaint will be checked by comparing the healthy side.
- Shoulder elastography on the non-hemiplegia side of patients: Patients over the age of 18 who apply to our clinic and have hemiplegia complaints will be evaluated. Patients' age, gender, occupation, habits, disease duration, upper extremity with complaints, dominant upper extremity, additional disease, weight and height values will be recorded. In the physical medicine and rehabilitation department examination of the patients, the patients will be evaluated with the brunnstrom staging used in hemiplegic patients. The elastography of the shoulder on the side with hemiplegia and the elastography of the shoulder on the side without complaints will be examined. Thus, the patient's side with the complaint will be checked by comparing the healthy side.

SUMMARY:
In our study, we aimed to examine the muscles and tendons of the shoulder region on the plegic side of patients with hemiplegia by elastography and to investigate whether there is a relationship between the course of the disease and the course of the lesions that will occur in the shoulder.

DETAILED DESCRIPTION:
Patients over the age of 18 who apply to our clinic and have hemiplegia complaints will be evaluated. Patients' age, gender, occupation, habits, disease duration, upper extremity with complaints, dominant upper extremity, additional disease, weight and height values will be recorded. In the physical medicine and rehabilitation department examination of the patients, the patients will be evaluated with the brunnstrom staging used in hemiplegic patients. The elastography of the shoulder on the side with hemiplegia and the elastography of the shoulder on the side without complaints will be examined. Thus, the patient's side with the complaint will be checked by comparing the healthy side.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer patients
2. Patients over 18 years old
3. Patients with hemiplegia
4. Patients without any rheumatic disease
5. Patients without any neurological deficit and muscle disease
6. Not having received ftr treatment to the shoulder area in the last 3 months
7. No injection to the shoulder area in the last 3 months
8. Not having any surgical procedure on the shoulder area
9. Not to be pregnant

Exclusion Criteria:

1. Patients with any rheumatic disease
2. Patients with any neurological deficit and muscle disease
3. To have received ftr treatment to the shoulder area in the last 3 months
4. Being under 18 years old
5. Having an infectious disease
6. Having any benign or malignant disease
7. Any surgical procedure to the shoulder area
8. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 who apply to our clinic and have hemiplegia complaints will be evaluated.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-05-05 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Shoulder Region With Share-Wave Ultrasound Elastography in Patients With Hemiplegia | 02/05/2023-02/05/2024
  Hemiplegia

CONTACTS AND LOCATIONS:
Locations (1):
- Harran University Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Şanlıurfa, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No